CLINICAL TRIAL: NCT02324166
Title: Cefazolin-Lidocaine Solution for Reducing Pain Associated With Subconjunctival Antibiotic Prophylaxis in Vitreo-Retinal Surgery
Brief Title: Cefazolin-Lidocaine Combination Solution to Reduce Antibiotic Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Wai-Ching Lam, Professor University of Toronto, Residency Program Director Dept. of Ophthalmology, Continuing Medical Education, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: CefazolinPain
Record Dates: First submitted 2014-12-18; First posted 2014-12-24 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-12

CONDITIONS: Vitreoretinal Surgery; Endophthalmitis
Keywords: cefazolin; lidocaine
MeSH Terms: conditions — Endophthalmitis | interventions — Cefazolin; Lidocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cefazolin (Active Comparator): For the control group, cefazolin will be drawn into a 1 mL syringe and 0.5 mL will be injected with a 30-gauge needle into the subconjunctival space. This will be performed at the end of the retinal surgery.
  Interventions: Drug: Cefazolin
- Cefazolin + Lidocaine (Active Comparator): For the comparator group, the cefazolin and 0.2 mL lidocaine 2% will be mixed together in the same 1 mL syringe and 0.5 mL of the mixed solution injected with a 30-gauge needle into the subconjunctival space. This will be performed at the end of the retinal surgery surgery.
  Interventions: Drug: Cefazolin; Drug: Lidocaine

INTERVENTIONS:
Drug: Cefazolin — cephalosporin antibiotic
Drug: Lidocaine — local anesthetic
  Arms: Cefazolin + Lidocaine

SUMMARY:
In retinal surgery, endophthalmitis is a sight-threatening eye infection that could complicate patient vision after the operation. At Toronto Western Hospital, for retinal surgery (operating at the back of the eye) it is common practice to administer an antibiotic (cefazolin) at the end of surgery, to reduce the risk of post-operative endophthalmitis. The antibiotic is administered by injection underneath the part of the eye called the conjunctiva. However, this antibiotic injection is often associated with high levels of post-operative pain. Previous studies have observed a reduction of this pain by injecting an anesthetic (lidocaine) in the subconjunctival space before the antibiotic. This study will seek to examine whether mixing 2% lidocaine with cefazolin before its injection will reduce post-operative pain in the retinal surgery setting.

DETAILED DESCRIPTION:
Endophthalmitis is a sight threatening eye infection that can complicate any type of intra-ocular surgery including vitreo-retinal surgery. The incidence, risk factors, management, microbiology and prognosis of endophthalmitis following vitreo-retinal surgery has been well described by a prospective international study, which demonstrated that this complication is quite rare but has a poor prognosis(1,2).

It is a common practice to administer antibiotic at the end of surgery(3), to reduce the risk of post-operative endophthalmitis. In Canada and Europe for anterior segment surgery, intracameral injection of an antibiotic is a common practice(4). In vitreo-retinal surgery, the anterior segment is often not breached, so rather than the antibiotic being delivered into the anterior chamber, it is administered by subconjunctival injection. However, such subconjunctival injection of antibiotic, such as cefuroxime (a second generation cephalosporin) is often associated with high levels of post-operative pain(5).

Local anesthesia for vitreo-retinal surgery is routinely achieved by either subtenon or retro-bulbar regional anaesthesia. Vitreo-retinal surgery at Toronto Western Hospital typically is performed with retro-bulbar anaesthesia, which involves the transcutaneous injection of anesthetic solution, often 2% lidocaine and 0.5% marcain, into the retrobulbar space using a needle6. At the end of surgery, subconjunctival cefazolin (Ancef) and steroid(Solucortef) are given, and surgeons have noticed that this often appears to cause discomfort in the end of surgery.

Although previous study has explored the reduction of pain through the use of buffered lidocaine injected in the subconjunctival space before cefuroxime for cataract surgery(5), the utility of mixing 2% lidocaine with cefazolin before subconjunctival injection has not yet been evaluated. This may serve as an effective method of lowering pain associated with cefazolin delivery in the retinal surgical setting.

ELIGIBILITY:
Inclusion Criteria:

* Patient is above the age of 18,
* Patient requires retinal surgery,
* Requires retro-bulbar anaesthesia for vitreo-retinal surgery,
* Patient is able to provide consent to the study

Exclusion Criteria:

* Patient is cognitively incapable of performing the study,
* Patient is unable to fully understand the study requirements and provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Score | 1 year
  The change in numerical pain scale scores pre-and-post sub-conjunctival cefazolin administration for patients either receiving cefazolin alone versus patients receiving a combination of cefazolin and 2% lidocaine.

CONTACTS AND LOCATIONS:
Overall Officials: Wai-Ching Lam, MD, Principal Investigator — University Health Network, Toronto

REFERENCES:
- [Background] Park JC, Ramasamy B, Shaw S, Prasad S, Ling RH. A prospective and nationwide study investigating endophthalmitis following pars plana vitrectomy: incidence and risk factors. Br J Ophthalmol. 2014 Apr;98(4):529-33. doi: 10.1136/bjophthalmol-2013-304485. Epub 2014 Jan 13. PMID 24420916
- [Background] Park JC, Ramasamy B, Shaw S, Ling RH, Prasad S. A prospective and nationwide study investigating endophthalmitis following pars plana vitrectomy: clinical presentation, microbiology, management and outcome. Br J Ophthalmol. 2014 Aug;98(8):1080-6. doi: 10.1136/bjophthalmol-2013-304486. Epub 2014 Mar 31. PMID 24686917
- [Background] Gower EW, Lindsley K, Nanji AA, Leyngold I, McDonnell PJ. Perioperative antibiotics for prevention of acute endophthalmitis after cataract surgery. Cochrane Database Syst Rev. 2013 Jul 15;7(7):CD006364. doi: 10.1002/14651858.CD006364.pub2. PMID 23857416
- [Background] Ong-Tone L, Bell A, Tan YY. Practice patterns of Canadian Ophthalmological Society members in cataract surgery: 2011 survey. Can J Ophthalmol. 2012 Apr;47(2):124-30. doi: 10.1016/j.jcjo.2012.01.012. PMID 22560416
- [Background] Kayarkar VV, Dinakaran S. Topical anesthesia for phacoemulsification and painless subconjunctival antibiotic injection. J Cataract Refract Surg. 2001 Feb;27(2):198-200. doi: 10.1016/s0886-3350(00)00564-2. PMID 11226781
- [Background] Lai MM, Lai JC, Lee WH, Huang JJ, Patel S, Ying HS, Melia M, Haller JA, Handa JT. Comparison of retrobulbar and sub-Tenon's capsule injection of local anesthetic in vitreoretinal surgery. Ophthalmology. 2005 Apr;112(4):574-9. doi: 10.1016/j.ophtha.2004.10.043. PMID 15808246
- [Background] Younger J, McCue R, Mackey S. Pain outcomes: a brief review of instruments and techniques. Curr Pain Headache Rep. 2009 Feb;13(1):39-43. doi: 10.1007/s11916-009-0009-x. PMID 19126370